CLINICAL TRIAL: NCT01809496
Title: Auditory Rehabilitation From the Perspective of the Significant Other
Brief Title: Hearing Aids, Counseling and the Significant Other
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: VA National Center for Rehabilitative Auditory Research (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, M. Samantha Lewis, Ph.D., Principal Investigator, VA National Center for Rehabilitative Auditory Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C7067W
Record Dates: First submitted 2013-03-06; First posted 2013-03-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aids; spouses; rehabilitation
MeSH Terms: conditions — Hearing Loss | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Informational counseling, patient only (Active Comparator): The purpose of this experimental group is to evaluate the effectiveness of informational counseling alone. This type of counseling is considered the standard of care in audiologic practice. Patients in this will review this material in detail with a member of the study team for approximately 30 minutes at the second visit. Spouses in this experimental group will be will review material regarding VA services with a member of the study team for about 30 minutes.
  Interventions: Behavioral: Informational Counseling
- Informational Counseling, couples (Experimental): The purpose of this experimental group is to evaluate the influence of spousal involvement when receiving informational counseling. In this manner, both patients and spouses are presented with the same information regarding hearing loss and hearing aids. Couples in this experimental group will be given the same information that the patients in the first group were given. At the second visit, couples in this group will review this information together with a member of the research team for approximately 30 minutes.
  Interventions: Behavioral: Informational Counseling
- Patient Centered Counseling,patient only (Experimental): In order to assess the effects of enhanced patient-centered counseling (PCC), the patients assigned to this group will meet together with either Dr. Lewis or the Research Audiologist for approximately 30 minutes of counseling. In addition to the PCC techniques used in audiology, this counseling also will involve the core components of motivational interviewing. These principles and methods will be used to allow the patient to clearly express his/her expectations of, concerns about, and motivations for hearing-aid use. The spouses in this experimental group will be given information regarding VA services. This material will be reviewed with a member of the research team for about 30 minutes at the second visit.
  Interventions: Behavioral: Patient Centered Counseling
- Patient Centered Counseling, couples (Experimental): In order to assess the influence of the spouse on the enhanced PCC process, the couples assigned to this group will meet together with either Dr. Lewis or the Research Audiologist for approximately 30 minutes of counseling. This counseling will be conducted with both the patient and the spouse together, giving both partners time to express their thoughts.
  Interventions: Behavioral: Patient Centered Counseling

INTERVENTIONS:
Behavioral: Informational Counseling
  Arms: Informational Counseling, couples; Informational counseling, patient only
Behavioral: Patient Centered Counseling
  Other Names: motivational interviewing
  Arms: Patient Centered Counseling, couples; Patient Centered Counseling,patient only

SUMMARY:
The purpose of this study is to examine the effect of enhanced patient-centered counseling (PCC) and the influence of spousal involvement in pre-fitting counseling on hearing-aid outcomes.

ELIGIBILITY:
Inclusion Criteria: Both men and women with hearing loss and their live-in partners will serve as subjects in this study. The subjects with hearing loss will have a mild to moderately-severe hearing loss in both of the ears, will have word recognition scores of 40% or better bilaterally, and will be about to get new hearing aids. Live-in partners may also have up to a moderately-severe degree of hearing loss but cannot have prior experience with hearing aids nor have plans to get hearing aids during the course of their participation in this study. Their word recognition scores should also be 40% or better bilaterally. All subjects also will meet the following additional inclusion criteria:

1. Age 20-85 years;
2. Intact mental status as assessed by the Mini-Mental State Examination (MMSE; Folstein, Folstein & McHugh, 1975);
3. No evidence of any major medical illness requiring long-term assistive care, as determined by the Katz Index of Independence in Activities of Daily Living (Katz, Down, Cash &Grotz, 1970);
4. Able to read and respond to English; and
5. Willing and able to give written informed consent to participate in this investigation.

Exclusion Criteria: Failure to satisfy any of the requirements listed above or if their live-in partner fails to meet the criteria.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
post-use subjective opinions regarding the hearing aids | 4-6 weeks after the hearing aid fitting
  questionnaires

SECONDARY OUTCOMES:
pre-use hearing aid expectations | immediately after the intervention at Visit #2 (Day 0)
  questionnaire

OTHER OUTCOMES:
self-efficacy | 4-6 weeks after the hearing aid fitting
  questionnaires
hearing aid use | 4-6 weeks after the hearing aid fitting
  datalogging

CONTACTS AND LOCATIONS:
Overall Officials: M. Samantha Lewis, PhD, Principal Investigator — VA National Center for Rehabilitative Auditory Research
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

REFERENCES:
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204